CLINICAL TRIAL: NCT00922220
Title: Immediate Effect of Physical Interventions for Low Back Pain
Brief Title: A Study of a Potential Mechanisms of Spinal Manipulation in the Treatment of Low Back Pain
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 343-2004
Record Dates: First submitted 2009-06-15; First posted 2009-06-17 (Estimated); Last update posted 2011-12-22 (Estimated); Status verified 2009-06

CONDITIONS: Low Back Pain
Keywords: low back pain; spinal manipulation; central sensitization; manual therapy
MeSH Terms: conditions — Low Back Pain | interventions — Manipulation, Spinal; Musculoskeletal Manipulations

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- stationary bike (Active Comparator): Participants rode a stationary bike for five minutes
  Interventions: Other: stationary bike
- lumbar extension exercises (Active Comparator): Participants performed four sets of fifteen lumbar extension exercises over five minutes
  Interventions: Other: lumbar extension exercise
- spinal manipulative therapy (Experimental): Participants received spinal manipulative therapy to the low back
  Interventions: Other: spinal manipulative therapy

INTERVENTIONS:
Other: stationary bike — Participants rode a stationary bike for five minutes
  Arms: stationary bike
Other: lumbar extension exercise — Participants performed four sets of fifteen lumbar extension exercises over fifteen minutes
  Other Names: press up
  Arms: lumbar extension exercises
Other: spinal manipulative therapy — participants received spinal manipulative therapy to the low back
  Other Names: spinal manipulation; manual therapy
  Arms: spinal manipulative therapy

SUMMARY:
The purpose of this study was to determine the immediate effect of 3 common physical therapy interventions for people experiencing low back pain on the perception of thermal pain. Additionally, the investigators wished to determine the influence of psychological factors related to fear and anxiety on their findings and to determine whether the effects of the individual interventions were local (specific to the area of application) or global (influenced regions away from the area of application).

ELIGIBILITY:
Inclusion Criteria:

* ages eighteen to sixty
* currently experiencing low back pain OR currently not experiencing low back pain and have not had an episode for the prior six months

Exclusion Criteria:

* non-English speaking
* systemic medical conditions (e.g. diabetes, hypertension)
* current use of psychiatric medication
* pregnancy
* signs and symptoms indicative of nerve root compression (reflex change, myotomal weakness, or sensation change)
* history of surgery to the low back

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 94 (Actual)
Dates: Start 2004-10; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Numeric Rating Scale | Prior to and immediately following assigned intervention

CONTACTS AND LOCATIONS:
Overall Officials: Steven Z George, Phd, Principal Investigator — University of Florida Department of Physical Therapy
Locations (1):
- University of Florida, Gainesville, Florida, United States

REFERENCES:
- [Result] George SZ, Bishop MD, Bialosky JE, Zeppieri G Jr, Robinson ME. Immediate effects of spinal manipulation on thermal pain sensitivity: an experimental study. BMC Musculoskelet Disord. 2006 Aug 15;7:68. doi: 10.1186/1471-2474-7-68. PMID 16911795
- [Result] Bialosky JE, Bishop MD, Robinson ME, Zeppieri G Jr, George SZ. Spinal manipulative therapy has an immediate effect on thermal pain sensitivity in people with low back pain: a randomized controlled trial. Phys Ther. 2009 Dec;89(12):1292-303. doi: 10.2522/ptj.20090058. Epub 2009 Oct 1. PMID 19797305